CLINICAL TRIAL: NCT04892147
Title: Movement-Oriented Behavioral Activation (MOBA) to Reduce Stationary Behavior
Brief Title: Movement-Oriented Behavioral Activation (MOBA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108020; 5P30AG064201 (NIH)
Record Dates: First submitted 2021-05-13; First posted 2021-05-19 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Wait-list control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Randomly selected to participate first in MOBA group
  Interventions: Behavioral: Mobility-Oriented Behavioral Activation
- Wait-list-control group (Other): Randomly selected for study assessments parallel with experimental group. Participates in MOBA after completion of the experimental group
  Interventions: Behavioral: Mobility-Oriented Behavioral Activation

INTERVENTIONS:
Behavioral: Mobility-Oriented Behavioral Activation — 12-weeks of mobility-oriented behavioral activation group

SUMMARY:
The purpose of this research study is to determine the acceptability, feasibility, and effectiveness of behavioral activation to increase everyday movement and reduce the amount of time spent daily in positions of prolonged standing and sitting. This intervention is call Movement-Oriented Behavioral Activation (MOBA). Participants will undergo a 60-minute screening that includes health and lifestyle questionnaires, mobility testing and a six-minute walk. Participants will complete the same procedures after completing MOBA. Each participant will be randomly assigned to an intervention group or a wait-list group. Both groups will participate in the same 12-week MOBA group protocol, but the intervention group participates first. During MOBA sessions, participants will set movement goals to reduce total time spent sitting and standing, and learn exercises and strategies to get more physical activity throughout the day and evening. At the end of the 12-week group, all participants, including those on the wait-list will be asked to complete the same questionnaires, mobility testing, and 6-minute walk as the beginning of the study. Total study duration for the intervention group is about 4 months. Total study duration for wait-list group will be about 8 months, which about half of that time spent in the waiting period.

Separate from the intervention there will be a focus group with prospective participants (N = 4-8) to collect information about physical activity perspectives and experiences to better align delivery of the intervention to the target cohort (participation in the focus group does not obligate participation in the intervention). A focus group will be conducted post intervention also. Participants enrolled in the intervention can participate in the focus groups.

DETAILED DESCRIPTION:
Overview. The study uses randomized waitlist-control design. We propose to randomly assign half of participants to (a) 10 weeks of MOBA intervention, and half of participants to (b) a 10-week waitlist, followed by 10 weeks of MOBA.

Intervention. MOBA is adapted from established protocols to integrate traditional behavioral activation (BA) principles with strategies to incorporate values-based, goal-directed movement into daily routines. The BA content of MOBA is adapted from co-investigator Dr. Smoski's intervention Behavioral Activation Therapy for Anhedonia (BATA). MOBA reduces depression-related content relative to BATA and increases focus on values that engage individuals in movement-related activity. MOBA is designed as a group intervention to leverage the reward value of social contact, and the positive influence of group problem-solving and accountability on behavior change. MOBA preserves the principles and general sequence of sessions used in BATA, but incorporates movement-oriented content: (a) provide psychoeducation about risks of physical inactivity, behavioral barriers to activity, and rationale for the treatment approach; (b) explore personal values, non-stationary, movement-oriented activities that support those values, and a hierarchical plan for goal attainment; (c) identify and assign weekly activities related to the valued goals; (d) address common barriers to engagement with valued activities including avoidance, low behavioral initiation, and an overemphasis on felt motivation as a prerequisite for action; and (e) monitor, support, and reward achieving behavioral goals. Content unique to MOBA includes: 1) demonstration and participation in physical activities that provide alternatives to stationary behavior, including select activities used in a previous study with the Dining Services cohort (e.g., stairs, body-weight squats, knee raises), and 2) generation of person-centered strategies for integrating movement-oriented activities into daily routines across the three domains of the Behavior Settings Model: 1) workplace sitting/prolonged standing, 2) screen-focused home activities, 3) time spent sitting in automobiles. Weeks 1-4 address topics a-c; weeks 5-12 address topics d-e. MOBA will be facilitated by a clinician (Dr. Potter) and a wellness educator (Dr. Tittle), who will be trained on the MOBA treatment manual. The facilitators' role is to provide teaching, support, encouragement, and guidance throughout the intervention. Weekly sessions will take place in a dedicated conference room near the workplace, during the last hour of the workday (4-5 pm), and is counted as paid time at work.

ELIGIBILITY:
Inclusion Criteria:

Pilot cohort will be composed of food service workers drawn employee by sponsor's organization. The age range was chosen to target the critical window for establishing the long-term geroprotective benefits of increasing movement-oriented behaviors. The workplace cohort was chosen because their work demands are characterized by a high level of stationary activity.

Exclusion Criteria:

1) individuals with moderate or greater depression severity (PHQ-9 > 14); and 2) individuals with significant mobility limitation, defined as inability to complete 6 Minute-Walk Test.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Potter, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pre-intervention focus group participants were not considered enrolled.
Groups:
- Experimental Group: Randomly selected to participate first in MOBA group
  Mobility-Oriented Behavioral Activation: 10-weeks of mobility-oriented behavioral activation group
- Wait-list-control Group: Randomly selected for study assessments parallel with experimental group. Participates in MOBA after completion of the experimental group
  Mobility-Oriented Behavioral Activation: 10-weeks of mobility-oriented behavioral activation group
Period: Overall Study
Arm/Group | Experimental Group | Wait-list-control Group
Started | 15 | 11
Completed | 13 | 11
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Wait-list-control Group | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.46 (6.75) | 55.27 (8.36) | 55.37 (7.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 11 | 22
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Movement-Oriented Behavioral Activation (MOBA)
Description: Survey questionnaire assessing participant experience of session content relevant to importance, competence achieved, enjoyment, activity change, group competition, and overall experience. Reported here is the mean response score on the Enjoyment scale, which surveyed 8 content topics on a 1-5 Likert scale, with higher values reflecting greater enjoyment (total range = 8-40). For the purposes of the analsyis, the mean of the Enjoyment scale was converted be comparable to original Likert scale range of 1-5, with a score of 3 characterizing the null hypotheis value of a "neutral" response.
Time Frame: Week 10 for the immediate intervention group, and Week 20 for the wait-list control group
Population: Participants from both groups who completed the questionnaire after their respective participation in the MOBA intervention. The a priori statistical plan was to examine acceptability ratings at end of intervention, which includes combining these data from both the experimental and waitlist groups for the reported analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Combined Experimental Group: Mobility-Oriented Behavioral Activation: 10-weeks of mobility-oriented behavioral activation group
Arm/Group | Combined Experimental Group
Number analyzed (Participants) | 22
score on a scale | 4.7 (0.4)
Statistical Analysis 1: Comparison: Combined Experimental Group; Test type: Other — Mean value of "Enjoyment" (8-item summed scale) tested against the value of a "Neutral" Likert response ("Neutral" value = 3); p < 0.001, t-test, 2 sided — The threshold for statistical significance was p = 0.05. The reported value is a calculated -p-value

2. Primary Outcome: Change in Short Physical Performance Battery (SPPB)
Description: The SPPB is a validated assessment of physical performance across three tasks: balance, gait speed, and chair stand. Each task is rated on a scale of 0-4, with a total range of range 0-12. Higher scores reflect better performance. Change = (Week 10 Score - Baseline Score).
Time Frame: Baseline, 10 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group | Wait-list-control Group
Number analyzed (Participants) | 13 | 11
units on a scale | -0.2 [-0.9 to 0.4] | -0.1 [-0.8 to 0.5]
Statistical Analysis 1: Comparison: Experimental Group vs Wait-list-control Group; Test type: Equivalence — Analyses were conducted using general linear models, controlling for baseline levels only with treatment group as the predictor of interest; p = 0.259, Regression, Linear — The threshold for statistical significance was p = 0.05

3. Primary Outcome: Change in Endurance as Measured by the 6-Minute Walk Test (6MWT)
Description: 6MWT is a validated measure of aerobic capacity/endurance as measured by the number of feet walked in six minutes following a specified route. A greater number of feet completed reflects greater aerobic capacity/endurance. Change = (Week 10 Score - Baseline Score).
Time Frame: Baseline, 10 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: feet walked in six minutes
Arm/Group | Experimental Group | Wait-list-control Group
Number analyzed (Participants) | 13 | 11
feet walked in six minutes | -39.9 [-229 to 150] | -87.5 [-267 to 92]
Statistical Analysis 1: Comparison: Experimental Group vs Wait-list-control Group; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.711, Regression, Linear — The threshold for statistical significance was p = 0.05

4. Secondary Outcome: Change in Behavioral Activation as Measured by the Behavioral Activation for Depression Scale (Short Form, BADS-SF).
Description: The BADs-SF is a validated short from of the original BADS. Both measures are self-report questionnaires designed to measures the mechanism of activation. The BADS-SF is composed of 9 items rated on a 0 to 6 scale. The total score range is 0-54, with higher scores reflecting greater engagement with rewarding activities. Change = (Week 10 Score - Baseline Score).
Time Frame: Baseline, 10 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group | Wait-list-control Group
Number analyzed (Participants) | 13 | 11
units on a scale | 2.6 [-0.9 to 6.2] | 5.8 [2.1 to 9.5]
Statistical Analysis 1: Comparison: Experimental Group vs Wait-list-control Group; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.214, Regression, Linear — The threshold for statistical significance was p = 0.05

5. Secondary Outcome: Change in Self-Reported Sedentary Time on the Past-day Adults' Sedentary Time Questionnaire (PAST)
Description: The Past-Day Adults' Sedentary Time questionnaire (PAST) is a validated questionnaire in which the participant estimates the is the hours spent sedentary across 7 domains of daily activity. The outcome variable was measured in total minutes converted to hours (minutes/60). Higher values represent more time spent sedentary. Change = (Week 10 Score - Baseline Score).
Time Frame: Baseline, 10 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: hours per day
Arm/Group | Experimental Group | Wait-list-control Group
Number analyzed (Participants) | 13 | 11
hours per day | -1.0 [-2.1 to 0.1] | -0.3 [-1.3 to 0.8]
Statistical Analysis 1: Comparison: Experimental Group vs Wait-list-control Group; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.317, Regression, Linear — The threshold for statistical significance was p = 0.05

6. Secondary Outcome: Change in Self-Reported Minutes of Moderate-to-Vigorous Physical Activity (MVPA)
Description: Self-reported minutes per week of moderate-to-vigorous physical activity. Moderate activity was calculated from number of days per week reported moderate physical activity (0-7) multiplied by average minutes reported per day. Vigorous physical activity calculated in the same manner. The total MVPA score was the sum of moderate and vigorous minutes reported. Greater number of minutes reflects higher levels of physical activity. Change = (Week 10 Score - Baseline Score).
Time Frame: Baseline, 10 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Experimental Group | Wait-list-control Group
Number analyzed (Participants) | 13 | 11
minutes per week | 78.4 [29.0 to 127.0] | 16.2 [-23.8 to 56.3]
Statistical Analysis 1: Comparison: Experimental Group vs Wait-list-control Group; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.056, Regression, Linear — The threshold for statistical significance was p = 0.05

7. Secondary Outcome: Change in Perceived Barriers to Activity
Description: The Barriers to Being Active Quiz has a score range from 0-63, with higher scores reflecting greater perceived barriers to activity.
Time Frame: Baseline, 10 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental Group | Wait-list-control Group
Number analyzed (Participants) | 13 | 11
score on a scale | 3.9 [-4.8 to 12.6] | 0.4 [-8.7 to 9.5]
Statistical Analysis 1: Comparison: Experimental Group vs Wait-list-control Group; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.562, Regression, Linear — The threshold for statistical significance was p = 0.05

ADVERSE EVENTS:
Time Frame: From enrollment until the conclusion of the 6-month program
Description: For the purposes of this study, an adverse event is defined as any undesired, noxious, or pathological change, as indicated by symptoms that occur in association with study participation. Pre-existing conditions that worsen during a study are considered AEs. Serious Adverse Events (SAE) are any adverse event that results in any of the following: Death or life-threatening illness including active suicidal ideation/attempt; Persistent or significant disability/incapacity; Hospitalization ≥24 hours
Arm/Group | Experimental Group | Wait-list-control Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT04892147/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT04892147/ICF_000.pdf